CLINICAL TRIAL: NCT02841072
Title: Chart Review Study of Medical Abortion at 64-70 Days of Gestation
Brief Title: Chart Review Study of Medical Abortion
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Other Study IDs: 1029
Record Dates: First submitted 2016-07-15; First posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Abortion, Medical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to document the rates of success and serious complications among women having outpatient medical abortions with 200 mg mifepristone + 800 buccal misoprostol at 64-70 days of gestation.

DETAILED DESCRIPTION:
The study will be conducted at US abortion clinics that have offered medical abortion with 200 mg mifepristone + 800 mcg buccal misoprostol to at least 20 women at 64-70 days of gestation. Designated staff at each site will review clinic records to identify and record data from every patient treated in that gestational week. Once data collection is completed, if the rate of success or serious complications at any clinic is substantially discordant from rates documented in the published literature, we may collect additional data on patients seeking medical abortion at 57-63 days, to aid in explaining results found in the 64-70 days group. In this situation, for each patient in the 64-70 days group, site staff will identify and record data from the next consecutive patient treated with this regimen at 57-63 days.

ELIGIBILITY:
Inclusion Criteria:

* Women at 64-70 days of gestation
* Received 200 mg mifepristone + 800 mcg buccal misoprostol for a medical abortion

Exclusion Criteria:

* Does not meet the inclusion criteria

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted at US abortion clinics that have offered medical abortion with 200 mg mifepristone + 800 mcg buccal misoprostol to at least 20 women at 64-70 days of gestation. Designated staff at each site will review clinic records to identify and record data from every patient treated in that gestational week.
Sampling Method: Non-Probability Sample
Enrollment: 579 (Actual)
Dates: Start 2015-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Abortion Success | 1 week
  Defined as a complete abortion without use of surgery
Serious complications | 1 month
  Defined as admission to hospital, receipt of parenteral antibiotics, surgery (laparoscopies, laparotomies, hysterectomies), transfusion, or death

SECONDARY OUTCOMES:
Proportion of ongoing pregnancies | 1 week
  Proportion of ongoing pregnancies after the initially dispensed mife-miso
Proportion of complete abortions without additional treatment | 1 week
  Proportion of complete abortions without additional treatment other than the initially dispensed mife-miso
Proportion of significant abortion complications | 1 month
  Proportion of significant abortion complications, including diagnosis of receipt of treatment for an abortion-related problem at an emergency department or urgent care center

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Raymond, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (2):
- United States (2):
  - Family Planning Associates- Northwest Chicago, Chicago, Illinois
  - Family Planning Associates- Downtown Chicago, Chicago, Illinois